CLINICAL TRIAL: NCT00158574
Title: Drug Options for Intermittent Preventive Treatment for Malaria in Infants in an Area With High Resistance to Sulfadoxine/Pyrimethamine: an Evaluation of Short and Long-acting Antimalarial Drugs
Brief Title: Kilimanjaro IPTi Drug Options Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Copenhagen (Other); National Institute for Medical Research, Tanzania (Other Government); Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: ITDCVF01
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: intermittent preventive treatment; malaria; efficacy; safety; drug options
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Mefloquine; chloroguanil, dapsone drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): IPTi placebo
  Interventions: Drug: Placebo
- Sulphadoxine-pyrimethamine (Experimental): IPTi SP
  Interventions: Drug: sulphadoxine-pyrimethamine; Drug: Sulphadoxine-pryrimethamine
- Mefloquine (Experimental)
  Interventions: Drug: mefloquine; Drug: IPTi mefloquine
- Chlorproguanil dapsone (Experimental)
  Interventions: Drug: Chlorproguanil-dapsone; Drug: Chlorproguanil dapsone

INTERVENTIONS:
Drug: sulphadoxine-pyrimethamine
  Other Names: Fansidar
  Arms: Sulphadoxine-pyrimethamine
Drug: mefloquine
  Other Names: Larium
  Arms: Mefloquine
Drug: Chlorproguanil-dapsone
  Other Names: Lapdap
  Arms: Chlorproguanil dapsone
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Sulphadoxine-pryrimethamine — IPTi doses 1 and 2, at ages 2 and 3 months, sulphadoxine 250mg, pyrimethamine 12.5mg IPTi doses 3, at 9 months of age, sulphadoxine 500mg, pyrimethamine 25mg
  Other Names: Fansidar
  Arms: Sulphadoxine-pyrimethamine
Drug: IPTi mefloquine — IPTi doses 1 & 2 at ages 2 & 3 months, mefloquine 125mg IPTi dose 3 at 9 months, mefloquine 250mg
  Other Names: Larium
  Arms: Mefloquine
Drug: Chlorproguanil dapsone — IPTi doses 1 and 2 at ages 2 and 3 months, doses 15mg chlorproguanil and 18.75mg dapsone IPTi dose 3 at 9 months of age, doses 22.5mg chlorproguanil and 28.13mg dapsone
  Other Names: Lapdap
  Arms: Chlorproguanil dapsone

SUMMARY:
Malaria and anaemia are major causes of morbidity and mortality in children in sub-Saharan Africa. Administration of three courses of sulfadoxine/pyrimethamine (SP) as intermittent preventive treatment (IPTi) to infants when they receive EPI vaccines reduced the incidence of malaria and anaemia in infants in an area with low SP resistance, low transmission pressure and high bednet use. However, it is not clear whether this observation can be generalised to areas with high transmission and high SP resistance. The mechanism of the protective effect of IPTi is unclear. There is an urgent need to identify other anti-malarial drugs that could be used for IPTi instead of SP.

This study objectives are:

1. Identification of a drug that could be used safely and effectively for IPTi instead of SP in areas, such as north eastern Tanzania, where there is a high level of resistance to SP and amodiaquine.
2. Determination of whether a short acting antimalarial drug (Lapdap) is as effective as a long acting drug (mefloquine) when used for IPTi.
3. Investigation of the effect of the intensity of transmission on the requirements for a long or short acting drug for IPTi.
4. Assessment of the effect of IPTi on the development of clinical immunity in children in low and high transmission areas.

A randomised trial with four treatment regimes is proposed which will be conducted in two different transmission settings. The four treatment regimens are as follows: (1) placebo; (2) mefloquine; (3) Lapdap; (4) SP. All medications will be given at the time of immunisation with DPT/polio 2, DPT/polio 3, and measles vaccines. The study will involve 1280 infants in a high endemic area and 2440 infants in a low endemic area, in Tanzania.The primary outcome is the incidence of clinical malaria.

DETAILED DESCRIPTION:
1. Study design

   The overall study design is a randomised trial of four treatment regimes in two different transmission settings. The four treatment regimes are as follows: (1) placebo, (2) mefloquine; (3) Lapdap; (4) SP. All medications will be given at the time of immunisation with DPT/polio 2, DPT/polio 3, and measles vaccines.
2. Study procedures

A list of study infants due for DPT/Polio 2 vaccination in each study EPI clinic on a given date will be generated from the enrolment database a week prior to the scheduled date.

When the study infants return for DPT& Polio 2 (contact 1) the following procedures will be carried out: (1) allocation of infants to one the four arms of the study; (2) administration of the first dose of the study drug and dispensation of the remaining two doses of drug to be given at home in the presence of a study field worker; (3) collection of blood samples for Hb, malaria parasite and blood spot for genetic markers of drug resistance parasites and haemoglobinopathies; (4) advice given to the caretakers to bring their children to the health facility if the child becomes ill before the next scheduled visit.

In both study areas, the first 200 children will be followed up on day 7 post-administration of IPTi first course (contact 1a) and a finger prick blood sample will be collected for determination of haemoglobin and preparation of blood film.

When the study infants return for DPT& Polio 3 (contact 2) the following procedures will be carried out: (1) administration of the first dose of the second course of the study drugs and dispensation of the remaining two doses of drugs to be given at home in the presence of a study field worker; (2) advice given to the caretakers to bring their children to the health facility if the child becomes ill before the next scheduled visit.

When the study infants return for measles (contact 3) the following procedures will be carried out: (1) administration of the first dose of the third course of the study drugs and dispensation of the remaining two doses of drugs to be given at home in the presence of a study field worker; (2) collection of blood samples for measles serology; (3) advice given to the caretakers to bring their children to the health facility if the child becomes ill.

In both study areas, the second 200 children will be followed up on day 7 post-administration of IPTi third course (contact 3a) and a finger prick blood sample will be collected for determination of haemoglobin and preparation of blood film.

A list of study infants who are due for blood examination one month after receiving course 3 of the study drugs will be generated from the contact3 database every month. These infants will be visited at home (contact 4) by a study team and a finger prick blood sample (400 μl) will be collected for determination of Hb, blood film preparation for malaria parasites and measuring anti-VSA antibodies. A random sample of 20% of infants will be visited at home at 11 months of age or two months after the 3rd course of the study drug (contact 5) and a finger prick blood sample will be collected for Hb and blood film preparation. Another random sample of 20% of children will be visited at home at 12 months of age or 3 months after the 3rd course of the drug (contact 6) and a finger prick blood will be collected for Hb and blood film preparation. Infant who had a blood sample taken at 11 months of age will be excluded from the sample of infants selected for collection of blood samples at 12 months of age. . All study children will be visited at home at the age of approximately 18 months (contact 7) and a finger prick blood sample (400 μl) will be obtained for determination of Hb, blood film preparation for malaria parasites and measuring anti-VSA antibodies.

All children will be visited at home at the age of approximately 24 months (contact 8) and finger prick blood sample will be obtained for screening for malaria using Optimal dipsticks and also for preparation of blood slides, filter paper samples and Hb. If a child is positive by dipstick test, is currently febrile (Temp >37.5° C) or has a history of fever within the past 2 days, and/or has a history of taking SP for a febrile illness during the previous week, the child will be treated with quinine.

If the dipstick test is positive for malaria and there is no history of fever within the past 2 days and no history of use of SP within the past week, the child will be given a full treatment course of any one of the three antimalarial drug used for IPTi ie SP, Lapdap or mefloquine, allocated randomly. The randomisation of treatment regime will be done in blocks of 6. Within each block of six envelopes, two will contain LapDap, two will contain MQ and Lapdap placebo for day 2 and 3, two will contain SP and Lapdap placebo for day 2 and 3. A random sample of 10% of children will be visited on day3 to assess whether the drugs were given to the children and a urine sample will be taken from approximately 200 children (selected randomly through out the year) for testing for mefloquine, dapsone and pyrimethamine using high performance liquid chromatography. All children who were treated with an antimalarial drug will be followed up on post treatment day 14 (contact 9) and on day 28 (contact 10). On these two visits a finger prick blood sample will be taken for examination of malaria parasite and filter paper sample obtained for subsequent determination of resistance markers to SP and Lapdap.

Randomisation and allocation of study groups

The unit of randomization will be an individual infant. Infants will be allocated to one of the study groups by permuted block randomization. Each study drug, including placebo, will be assigned 4 group codes; there will be 16 study groups in total in each study site and these will be colour coded. An independent statistician (Dr Tom Smith) will prepare the randomization scheme during the preparatory phase of the study. 233 blocks of 16 blister packs of study drugs [80 blocks (1280/16 = 80) for the high transmission area, and 153 blocks (2448/16 = 153) for the low transmission area] will be prepared and the study drug codes will be kept by the independent statistician.

The tablets will be crushed and mixed with syrup at the time of administration. The first dose will be administered at the EPI clinic by a designated member of the study team. The drugs for day 2 and 3 will be dispensed in blister packs and the caretakers will be advised to administer the drugs at home. The level of compliance and side effects of the drug will be monitored by the compliance assessment team during home visits made on day 2 and day 3. If drugs had not been given by the caretakers, the project staff will administer the drugs with the consent of the caretaker.

Oral administration of mefloquine can induce vomiting in children suffering from clinical malaria. We will observe the incidence of vomiting over an initial period of three months and report this information to the Data, Safety and Monitoring Board (DSMB). If the incidence of vomiting is significant, the DSMB may recommend that the schedule of mefloquine administration should be changed to a split dose (15 mg /kg on day 1 and 10 mg/kg on day 2).

Monitoring compliance and safety

Compliance with the three days of medication will be assessed by field staff during their visits on days 2 and 3. Urine samples will be collected on a random basis throughout the course of the trial at the day 3 visit and tested for mefloquine, dapsone and pyrimethamine using high performance liquid chromatography (HPLC).

Determining the safety and acceptability of mefloquine and Lapdap when used for IPTi will be a major objective of the study. This will be accomplished in three main ways:

1. Changes in haemoglobin during the week following treatment will be measured and related to the presence or absence of parasitaemia and or fever at the time of treatment. Data for each of the 16 treatment groups will be collated by the investigators and given to the DSMB which will be asked to break the code for these subjects and to determine if there is are any concerns over a fall in Hb in the approximately 200 infants who have received Lapdap. It will be possible to compare findings in these children with those children who receive mefloquine, SP or placebo. If necessary, the G-6-P-D status will be determined in any children who show a drop in Hb and in matched controls.
2. . At the time of the day 3 follow-up, a questionnaire will be completed which asks about the health of the infant since the time of drug administration.
3. . An adverse events reporting system will be established in each of the health centres participating in the trial. Any severe adverse event will be reported to the chair of the DSMB and to GSK within 48 hours.

Drugs used for IPTi must not have any suppressive on the immune response to EPI vaccines given concurrently. An impact on measles vaccination is the issue of most concern. Therefore, a serum sample will be collected at the age of 9 months before administering measles vaccination and one month after the administration of the vaccine. Antibody concentrations to DPT antigens may be measured in these samples.

Surveillance of clinical malaria

All study infants will be encouraged to attend the study health facilities for any illness. At these visits a health questionnaire will be completed and temperature recorded using an electronic thermometer. A finger prick blood sample will be collected for Hb and malaria parasite and for detection of molecular markers of resistance from all infants attending the study health facilities for any illness that is clinically diagnosed as malaria.

Children with proven or presumptive malaria will be treated with quinine according to the MoH guidelines for managing treatment failures following first line drugs.

To ensure that IPTi with any of the study drugs does not lead to a rebound in the incidence of severe malaria or anaemia during the second year of life all infants enrolled in the study will be followed until they reach the age of 24 months. During their second year of life, all episodes of possible malaria or anaemia in infants who present to health centre in the study area will be documented.

Monitoring of the trial

The trial will be conducted under conditions of good clinical practice (GCP), following as closely as possible the ICH guidelines. Standard operating procedures (SOPs) will be developed for all major operations. A DSMB will be established to look after the trial. Discussions will be held with the DSMB prior to the start of the trial to identify their requirements for adverse events reporting and these will be met. The DSMB will also be consulted about the advisability of an interim analysis, in particular for the SP group as this drug may prove to be ineffective.

At each study site, a local physician will be assigned to be the local safety monitor. In the event of a serious adverse event associated with a study drug, the local safety monitor will be empowered to break the code for that child and, if it is considered necessary to temporarily suspend the trial, prior to discussion with the DSMB.

It is proposed that a clinical monitor will be appointed by the IPTi consortium to monitor all the trials conducted under its auspices and it is anticipated that the monitor will visit the study site on at least one occasion during the trial and provide advice that will help to ensure that the study is conducted to the highest clinical standard.

ELIGIBILITY:
Inclusion Criteria:

* All infants attending EPI clinics at the 12 study health facilities for first vaccinations. Infants who live within the catchment area of the study health facility and are less than 3 months of age at the time of DPT and Polio 1 vaccination will be eligible for inclusion in the study.

Exclusion Criteria:

* Infants having any of the following conditions will be excluded: (1) history of allergy to study drugs; (2) history of convulsions; (3) clinical features of severe malnutrition or chronic illness including infants with signs of AIDS [HIV prevalence in women of reproductive age in the study area was 11.5% in 1999]39 (4) plans to leave the study area before 12 months of age.(5) weighs <4.5 kgs (6) caretaker declines to give consent.

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2419 (Actual)
Dates: Start 2005-01; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
1. Incidence of clinical malaria: [(history of fever during previous 2 days or axillary temperature >37.5ºC) + parasitaemia of any density + absence of any other obvious causes of fever] during the period of 3-11 months of age | 3-11 months of age

SECONDARY OUTCOMES:
1.Mean Hb at 10-12 months of age (one month after the third course of IPTi) | 10-12 months of age
2.Incidence of severe anaemia (Hb <7 g/dl) during the period of 3-11 months of age | 3-11 months of age
3.Prevalence of parasitaemia at 10-12 months of age (one month after the third course of IPTi) | 10-12 months of age
4.Incidence of clinical malaria [as defined above] during the period of 12-23 months of age. | 12-23 months of age
5.Level and repertoires of plasma antibodies to Plasmodium falciparum variant surface antigen (anti-VSA antibodies) at 10 and 18 months of age. | 10 and 18 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Roly Gosling, MBChB, MRCP, Study Director — London School of Hygiene and Tropical Medicine; Daniel Chandramohan, MBBS,PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Brian Greenwood, FRCP, FRS, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Ministry of Health, Korogwe and Same District MCH clinics, Tanga, Tanga and Kilimanjaro, Tanzania

REFERENCES:
- [Derived] Cairns M, Gosling R, Carneiro I, Gesase S, Mosha JF, Hashim R, Kaur H, Lemnge M, Mosha FW, Greenwood B, Chandramohan D. Duration of protection against clinical malaria provided by three regimens of intermittent preventive treatment in Tanzanian infants. PLoS One. 2010 Mar 1;5(3):e9467. doi: 10.1371/journal.pone.0009467. PMID 20209126
- [Derived] Gosling RD, Gesase S, Mosha JF, Carneiro I, Hashim R, Lemnge M, Mosha FW, Greenwood B, Chandramohan D. Protective efficacy and safety of three antimalarial regimens for intermittent preventive treatment for malaria in infants: a randomised, double-blind, placebo-controlled trial. Lancet. 2009 Oct 31;374(9700):1521-32. doi: 10.1016/S0140-6736(09)60997-1. Epub 2009 Sep 16. PMID 19765815